CLINICAL TRIAL: NCT07102147
Title: Increasing Adoption of a Telehealth-Delivered Collaborative Care Program for Patients With Lung Cancer: A Pilot Study
Brief Title: Telehealth Collaborative Care Model (CoCM) in Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexandria Muench, Staff Psychologist, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPCC 31524; P50CA271338 (NIH); 857520 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2025-07-18; First posted 2025-08-03 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer (Diagnosis); Anxiety; Depression in Adults
Keywords: Lung cancer; Anxiety; Depression; Collaborative care
MeSH Terms: conditions — Lung Neoplasms; Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Touch Outreach (Experimental): Patients in the high touch outreach arm will receive a gain-framed message via text (preferred modality), MyPennMedicine message, email, and/or postal mail that links to the digital screener; an informational flyer about collaborative care sent via postal mail, the MyPennMedicine portal, email, and/or text; and a direct request from their oncology provider to collaborative care for those patients who have not responded to outreach efforts by their next oncology visit post-referral.
  Interventions: Behavioral: High Touch Outreach
- Standard Outreach (No Intervention): Patients in the standard outreach arm will receive a standard message sent via text (preferred modality), MyPennMedicine message, email, and/or postal mail that links to the digital screener; this message is one that is similar to that already used in Penn Integrated Care's practice.

INTERVENTIONS:
Behavioral: High Touch Outreach — Gain-framed message, informational flyer, and direct request
  Arms: High Touch Outreach

SUMMARY:
The goal of this trial is to compare the impact of two outreach strategies (high touch vs. standard outreach) on a collaborative care program delivered via telehealth to patients with lung cancer.

DETAILED DESCRIPTION:
The goal of this project is to pilot test the effectiveness of using a more-intensive (high touch) outreach strategy to increase the reach of an adapted, standard of care CoCM for patients with lung cancer who are experiencing depression and/or anxiety. The investigators will specifically test the effect of two outreach strategies (high touch vs. standard outreach) on reach of the CoCM program (primary outcome) and on several secondary implementation and effectiveness outcomes. Given the demonstrated efficacy of the CoCM in patients with cancer, the main target of this research study is the impact of the outreach strategies and delivery of the CoCM via telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 years or older.
* Are currently being seen by Penn Medicine Thoracic Oncology for lung cancer treatment or survivorship care.
* Are referred to collaborative care by a Penn Medicine Thoracic Oncology clinician for treatment of depression, anxiety, or other psycho-therapy services.

Exclusion Criteria:

* Are already receiving psycho-therapy treatment services outside of Penn Medicine's collaborative care program, Penn Integrated Care (PIC).
* Have a significant and/or untreated medical and/or psychiatric co-morbidity (e.g., other cancers, schizophrenia, acute suicidal and/or homicidal ideation) that make them ineligible for the Penn CoCM program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Reach - Completion of the intake assessment amongst referred patients. | Measured per patient up to 30 days after randomization.
  The number of referred patients that complete the intake assessment divided by the total number of referred patients.

SECONDARY OUTCOMES:
Treatment Initiation - Completion of one or more oncology-based collaborative care appointments amongst patients deemed to be appropriate for oncology-based collaborative care at intake. | Measured per patient up to 60 days after randomization.
  The number of patients deemed to be appropriate for the oncology-based CoCM at intake who go on to complete one or more oncology-based CoCM appointments divided by the total number of patients deemed to be appropriate for the oncology-based CoCM at intake.
Treatment Retention - Completion of oncology-based collaborative care appointments amongst patients deemed to be appropriate for oncology-based collaborative care at intake. | Measured per patient at end of collaborative care treatment (assessed up to 6 months).
  Number of oncology-based collaborative care appointments completed amongst patients deemed to be appropriate for the oncology-based CoCM at intake.
Clinical Effectiveness (PHQ-9) - Change in symptom measure using the Patient Health Questionnaire-9 (PHQ-9) validated instrument. | Measured per patient at first collaborative care appointment (baseline) and at end of collaborative care treatment (up to 6 months).
  The change in PHQ-9 score from the patient's collaborative care intake appointment to the appointment most proximal to the patient's discharge. The instrument's minimum value is 0 and maximum value is 27, with a higher score indicating a worse outcome.
Clinical Effectiveness (GAD-7) - Change in symptom measure using the Generalized Anxiety Disorder-7 item (GAD-7) validated instrument. | Measured per patient at first collaborative care appointment (baseline) and at end of collaborative care treatment (up to 6 months).
  The change in GAD-7 score from the patient's collaborative care intake appointment to the appointment most proximal to the patient's discharge. The instrument's minimum value is 0 and maximum value is 21, with a higher score indicating a worse outcome.
Clinical Effectiveness (PROMIS Fatigue) - Change in symptom measure using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form 7a validated instrument. | Measured per patient at first collaborative care appointment (baseline) and at end of collaborative care treatment (up to 6 months).
  The change in PROMIS Fatigue - Short Form 7a score from the patient's collaborative care intake appointment to the appointment most proximal to the patient's discharge. The instrument's minimum value is 7 and maximum value is 35, with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria Muench, PsyD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No